CLINICAL TRIAL: NCT04601376
Title: To Implement and Test the Mobile Monitoring Tool to Identify SSI (R33 Phase)
Brief Title: Testing of Mobile Monitoring System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robin Kamal, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 57543
Record Dates: First submitted 2020-09-08; First posted 2020-10-23 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mobile monitoring group (Experimental)
  Interventions: Behavioral: Mobile Monitoring Tool

INTERVENTIONS:
Behavioral: Mobile Monitoring Tool — a text-messaged based outcomes collection system

SUMMARY:
We will complete a prospective, observational study comparing the accuracy of the mobile monitoring tool on identifying SSI compared to manual review.

ELIGIBILITY:
Inclusion Criteria:

* Orthopaedic surgery patient at hospital 175

Exclusion Criteria:

* no access to mobile phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Promis PF Short form (change in self reported capability) | 1 day, 1 week, 2 week, 4 week, 12 weeks after surgery
  PROMIS Physical Function instruments measure self-reported capability rather than actual performance of physical activities. It is scored from 0-100, a higher score indicates better physical function

IPD SHARING:
Plan to Share IPD: No